CLINICAL TRIAL: NCT04797988
Title: Eon® Flanks Safety Clinical Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominion Aesthetic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0000000160
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- eon FR 1064 nm Device (Experimental): Patient will be treated with the eon FR 1064 nm device.
  Interventions: Device: eon® FR 1064 nm device

INTERVENTIONS:
Device: eon® FR 1064 nm device — The subject will be treatment area - flanks, will be treated with the eon device.

SUMMARY:
This study is designed to provide objective evidence regarding the safety of eon® treatment of the flanks.

DETAILED DESCRIPTION:
This study is designed to provide objective evidence regarding the safety of eon® treatment of the flanks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female > 18 years or older seeking treatment for unwanted fat in the flanks.

  * Subject must be able to read, understand and sign the Informed Consent Form (ICF) in English.
  * Subject has sufficient thickness (≥ 20 mm) of adipose tissue on the flanks area.
  * Subject must be willing and able to adhere to the treatment and follow-up visit schedule.
  * Subject is willing to have photographs and ultrasound measurements taken of the treated area.
  * Female subjects must be using medically acceptable form of birth control during the entire course of the study or may be post-menopausal, or surgically sterilized.

Exclusion Criteria:

* • Subject had an aesthetic fat reduction procedure in the treatment area within the previous year

  * Subject was pregnant in the last 3 months, intending to become pregnant, postpartum or nursing in last 6 months
  * Subject has an infection, dermatitis or a rash in the treatment area.
  * Subject has tattoos or jewelry in the treatment area or within the treatment area site or photography frame.
  * Subject has a history of keloid scarring, hypertrophic scarring or of abnormal wound healing.
  * Subject has a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
  * Subject has a history of a known bleeding disorder.
  * Subject has a known photosensitivity to the study laser wavelength, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
  * Subject has known collagen, vascular disease or scleroderma.
  * Subject has undergone a surgery or procedure in the treatment area within 6 months of treatment, which is still healing.
  * Subject suffers from significant concurrent illness, such as insulin-dependent diabetes, peripheral vascular disease or peripheral neuropathy.
  * Subject is undergoing systemic chemotherapy for the treatment of cancer.
  * Subject is using gold therapy for disorders such as rheumatologic disease or lupus.
  * Subject has participated in a study of another device or drug within three months prior to enrollment or during the study.
  * As per the investigator's discretion, the subject has any physical or mental condition which might make it unsafe for the subject to participate in this study.
  * Subject has ongoing use of steroids or secondary rheumatoid drugs.
  * Subject is actively taking psychotropic medications.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation eon® treatment of the flanks (Adverse Events) | 2 weeks
  Adverse Events will be assessed to include ultrasound evaluations with a single expert sonographer identifying the pre-treatment versus Week 2 post-treatment.

SECONDARY OUTCOMES:
Subject Satisfaction | 2 weeks
  Subject Questionnaires will be completed by subjects at the end of the study to determine subject satisfaction with the procedure. Subjects will respond using a scale of 1-6, with 1 being extremely satisfied and 6 being extremely dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Fiala Aesthetics, Altamonte Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiala T, Lavin P. Safety of a 1064-nm robotic laser system for noninvasive lipolysis of the flanks. Lasers Surg Med. 2022 Jul;54(5):672-681. doi: 10.1002/lsm.23532. Epub 2022 Mar 9. PMID 35266172